CLINICAL TRIAL: NCT05639348
Title: Validation of a Risk Assessment Model for Postoperative Delirium Based on Artificial Intelligence
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Innosuisse - Swiss Innovation Agency (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-00990; am21Dell- Kuster
Record Dates: First submitted 2022-11-23; First posted 2022-12-06 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Postoperative Delirium (POD)
Keywords: Perioperative neurocognitive disorders (PND); Postoperative cognitive dysfunction (POCD); Acute neuropsychiatric disorder; Cognitive testing; Artificial intelligence (AI)-based algorithm PIPRA; Intensive Care Delirium Screening Checklist (ICDSC); 4 "A" Tests (4AT)
MeSH Terms: conditions — Emergence Delirium; Postoperative Cognitive Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection on POD for calculation of the PIPRA score — Data collection for presence of POD as diagnosed by the 4 "A" Tests (4AT) or the Intensive Care Delirium Screening Checklist (ICDSC). The collected data will be used to validate the existing PIPRA algorithm and to improve the algorithm and evaluate it in a cross-validation setting. For the model validation the area under the receiver operating characteristics (ROC) curve (AUC) will be computed.

SUMMARY:
Postoperative delirium (POD) is a frequent postoperative complication in the elderly, characterised by fluctuating disturbances in attention, awareness, and cognition. Identifying the patients at highest risk of developing POD was the aim of the artificial intelligence (AI)-based algorithm PIPRA. This prospective cohort study is to externally validate the AI-based PIPRA algorithm. The primary endpoint is the performance (AUC) of the PIPRA algorithm in predicting POD. The secondary endpoint is the performance (AUC) of the clinicians in predicting POD (and how it compares with the performance of the PIPRA algorithm).

DETAILED DESCRIPTION:
Perioperative neurocognitive disorders (PND) include postoperative delirium (POD) and postoperative neurocognitive disorder or postoperative cognitive dysfunction (POCD). POD is recognised as a frequent postoperative complication in the elderly, occurring in 10% to 50% of older patients after major surgical procedures. POD usually occurs in the early postoperative period and is defined as an acute neuropsychiatric disorder. It is characterised by fluctuating disturbances in attention, awareness, and cognition. The American Society of Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Postoperative Delirium Prevention recommend focusing on identifying those patients at highest risk of developing POD. Identifying these highest risk patients was the aim of the artificial intelligence (AI)-based algorithm PIPRA, which was created based on an individual participant data (IPD) meta-analysis including more than 2500 patients. This risk-prediction algorithm uses standard data (i.e. age, height, weight, history of delirium, cognitive impairment, ASA status, number of medications, preoperative C reactive protein (CRP), surgical risk and laparotomy), which are routinely collected before surgery. PIPRA was internally validated with an area under the curve (AUC) of 0.837 with 95% confidence interval 0.808 to 0.865, when plotting the true positive rate against the false positive rate. The aim of this prospective cohort study is to externally validate the AI-based PIPRA algorithm.

First, the anaesthesiologist in charge will be asked to evaluate, based on his/her experience (quantified in years of anaesthesia practice), the risk for the included patient to develop POD (categorised as low, intermediate, high or very high). Next, an investigator will assess included patents in a systematic and reproductible manner. After surgery, an investigator will visit the patient twice daily from postoperative day 1 to 5 or until hospital discharge (whichever occurs first) to screen for delirium using the 4AT or the ICDSC. The PIPRA score will be calculated separately by the coordinating study centre.

ELIGIBILITY:
Inclusion Criteria:

* Surgical patients ≥60 years old
* Planned postoperative hospital stay ≥ 2 days
* Consent from patient

Exclusion Criteria:

* Preoperative delirium
* Insufficient knowledge in German or French
* Intracranial surgery
* Cardiac surgery
* Surgery within the two previous weeks
* Patient unable to consent

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive surgical patients at multiple sites in Switzerland.
Sampling Method: Probability Sample
Enrollment: 993 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Change in 4 'A's Test (4AT) to evaluate presence of POD | Twice daily (morning and evening) from postoperative day 1 until postoperative day 5, hospital discharge or a positive diagnosis of POD, whichever occurs first.
  4 'A's Test (4AT) is a bedside medical scale with 4 parameters:
  1. Alertness
  2. Abbreviated mental test-4 (AMT4)
  3. Attention (months backwards test)
  4. Acute change or fluctuating course. The score range is 0-12, with scores of 4 or more suggesting possible delirium. Scores of 1-3 suggest possible cognitive impairment.
Change in Intensive Care Delirium Screening Checklist (ICDSC) to evaluate presence of POD | Twice daily (morning and evening) from postoperative day 1 until postoperative day 5, hospital discharge or a positive diagnosis of POD, whichever occurs first.
  The ICDSC is an 8-item delirium screening instrument (range: 0-8 points) that evaluates a patient's level of consciousness, inattention, disorientation, hallucinations or delusions, psychomotor activity, inappropriate speech or mood, sleep disturbance and fluctuation of symptoms (no delirium with a score of 0, less than clinical threshold symptoms of delirium with a score of 1-3 and clinical delirium with a score of 4-8).

CONTACTS AND LOCATIONS:
Overall Officials: Luzius Steiner, Prof. Dr. med., Principal Investigator — University Hospital Basel, Department of Anaesthesiology
Locations (3):
- Switzerland (3):
  - University Hospital Basel, Anaesthesiology, Basel
  - Hôpitaux Universitaires de Genève, Anesthesiology, Geneva
  - Centre Hospitalier Universitaire Vaudois, Anesthesiology, Lausanne